CLINICAL TRIAL: NCT05833854
Title: The Effect of Use of Virtual Reality Glasses and Manual Pressure Method on the Level of Pain and Fear in Children During Intramuscular Injection
Brief Title: The Effect of Two Different Methods Applied During Intramuscular Injection on the Level of Pain and Fear in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selmin Kose (Other)
Responsible Party: Sponsor-Investigator, Selmin Kose, Associate Professor Doctor, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 732202
Record Dates: First submitted 2023-04-02; First posted 2023-04-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Intramuscular Injection
Keywords: manual pressure; virtual reality glasses; intramuscular injection; pain; fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality glasses group (Experimental): The study group (n=25) will watch a video with virtual reality glasses during the intramuscular injection.
  Interventions: Other: Virtual reality glasses group
- Manual pressure group (Experimental): In the study group (n=25), pressure will be applied to the area to be injected for 10 seconds before the intramuscular injection procedure.
  Interventions: Other: Manual pressure group
- Control group (No Intervention): The control group (n=25) will not be subjected to any application other than intramuscular injection, which is routinely applied in pediatric emergency.

INTERVENTIONS:
Other: Virtual reality glasses group — It is suggested that the use of virtual reality glasses during the injection will positively affect the pain and fear levels in children who received penicillin injection in the pediatric emergency department where the study was conducted.
  Arms: Virtual reality glasses group
Other: Manual pressure group — In the pediatric emergency department where the study was conducted, pressure will be applied to the area to be injected for 10 seconds before the injection procedure in children who received penicillin injection. Pressing with the thumb of the hand, which will be passive in the pressing application, will be understood by the whitening of the nail, and thus pressure will be applied to the skin. It is suggested that it can positively affect pain and fear levels.
  Arms: Manual pressure group

SUMMARY:
This study was planned to determine the effects of using virtual reality glasses and manual pressure during intramuscular injection on the level of pain and fear in children. The study will consist of children aged 6-10 years who come to the Pediatric Emergency Service injection room for prescription penicillin injection and meet the inclusion criteria. One of the main purposes of nursing care is to relieve the child's pain and improve the quality of life. In this context, it has been suggested that two different methods used by the researcher can positively affect the levels of pain and fear. For this reason, it is aimed to determine the efficiency level of two different methods.

DETAILED DESCRIPTION:
75 children and parents meeting the inclusion criteria will be included in the study. For the penicillin injection prescribed by the doctor, the child and the parent who come to the pediatric emergency injection room of the hospital where the research is carried out are informed about the study and the parent is asked to sign the "Informed Consent Form". . After obtaining the consent of the family, the "Child-Parent Information Form" is filled by the researcher through the parent. Simple randomization will be done to give an equal number of samples to the control, virtual reality glasses and manual pressure group to be applied to the child who will participate in the study. Randomization of the study will be done with the online program at the URL https://www.randomizer.org/. Children to be included in the sample will be divided into three groups by randomization method. The numbers from 1 to 75 will be entered into the program without repeating, in order to determine which group the children included in the study will be in. The children who will form the study group through the program will be randomly distributed into 3 groups. . The two interventions in the study will be virtual reality glasses (n=25) and manual pressure (n=25) and control group (n=25).

In the control group (n=25), the child, the parent and the researcher will evaluate the children's fear levels before the procedure with the Child Fear Scale. In this group, a routine intramuscular injection will be made into the vastus lateralis muscle and the researcher will perform the application. No intervention other than routine will be applied. After the intramuscular injection, the pain level of the children will be evaluated by the child, the parent and the researcher with the Facial Expressions Pain Scale-Remodeled.

The group (n=25) wearing VR Glasses will be shown an age-appropriate VR video alongside the routine practice. Before the procedure, the level of fear will be evaluated as in the control group. A virtual reality VR video is watched 1 minute before the intramuscular injection. The child who continues to watch the video is placed on his back and penicillin is injected intramuscularly into the vastus lateralis muscle. Post-injection pain level will be evaluated as in the control group. Virtual reality glasses compatible with "VR BOX 3D" smartphones will be used in this group. Product weight: 0.414 kg. Product size (length x depth x height): 19.5 x 14 x 11 cm/ 7.66 x x5.50 x 4.32 inches. No power adapter or connection cable other than the phone will be needed during use. All children participating in the research will watch the "Hidden Underwater World", which is recommended by taking the opinion of an expert (child developmentist) suitable for their age. The virtual reality glasses used in the application will be disinfected and ready for the next application.

The manual pressure group (n=25) will be evaluated with the Child Fear Scale before the procedure. In addition to the routine application, pressure will be applied to the area to be injected for 10 seconds before the injection process. Pressing with the thumb of the hand, which will be passive in the pressing application, will be understood by the whitening of the nail, and thus pressure will be applied to the skin. Then, as in other groups, an injection will be made into the vastus lateralis area. After the injection, the child will be evaluated in terms of pain with the Facial Expressions Pain Scale revised by the parent and the researcher.

Informed Consent Form, Child-Parent Information Form, Child Fear Scale and Facial Expressions Pain Scale-Revised will be filled for each child who will participate in the study. It is planned to fill the Child Fear Scale before the injection and the Facial Expressions Pain Scale-Revised after the injection.

It is planned that the scales to be applied to the child and parent who will participate in the research will be applied face to face in the injection room of the hospital and 10-15 minutes will be given for each application.

The obtained data will be evaluated using the necessary statistical tests in the computer environment. Evaluation methods will be chosen based on whether the data is homogeneously distributed. If it has a homogeneous distribution, parametric tests will be used. If it does not have a homogeneous distribution, non-parametric methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to the pediatric emergency service for the administration of a penicillin antibiotic group drug,
* Absence of a significant chronic disease,
* Absence of visual and auditory disabilities,
* Having no communication problems and being conscious,
* No previous history of fainting during injection,
* Not taking analgesics in the last three hours,
* Percentile value is in the range of 3-97 points,
* Injection into the vastus lateralis muscle can be applied,
* The child's and parent's willingness to participate in the research.

Exclusion Criteria:

* The percentile value is below 3 and the percentile value is above 97,
* Family's inability to cooperate in the assessment of pain and fear,
* Having a diagnosed physical or mental disability,
* To have taken analgesics in the last 3 hours,
* Presence of incision and scar tissue in the area to be injected,
* The child's and parent's refusal to participate in the research.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale | The child's fear level will be evaluated by 3 people (child, parent and researcher) 2 minutes before intramuscular penicillin injection is given to the whole group. This process will take 1 minute.
  The purpose of the Child Fear Scale is to evaluate the fear level of children. It consisted of five facial expressions ranging from neutral expression (0 = No anxiety) to fearful expression (4 = Severe anxiety).

SECONDARY OUTCOMES:
Facial Expressions Pain Scale-Revised | Two minutes after intramuscular penicillin injection is given to the whole group, the child's pain will be evaluated by 3 people (child, parent and researcher). This process takes 1 minute.
  It is a valid and reliable scale that children can express themselves in their painful situations. It consists of 6 facial expressions that determine the severity and presence of pain by scoring between 0 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE KURTAR, RN, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Selmin Köse, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to Hospital policy, the individual participant data can not be shared with anyone except researchers.

REFERENCES:
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/24134180/